CLINICAL TRIAL: NCT05777382
Title: Quality of Life of Postnatal Mothers Attending Maternal and Child Health Clinic in Biratnagar
Acronym: QoL
Status: Completed | Type: Observational
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Pratiksha Chapagain, Principal Investigator, Tribhuvan University, Nepal
Other Study IDs: 131(6-N-E)2/075/076
Record Dates: First submitted 2023-02-18; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: inquiry to postnatal mothers — structured questionnaires was asked to postnatal mothers

SUMMARY:
Objectives: Assessing health-related quality of life (HRQoL) and its predictors is essential for providing adequate healthcare and developing necessary interventions in women post-delivery. This study intended to determine the HRQoL score and predictors among women post-delivery in Nepal.

Methodology: This was a cross-sectional study using non-probability sampling conducted at the Maternal and Child Health (MCH) Clinic of Koshi Hospital, Province 1, Nepal. The study participants were 129 women post-delivery to 12 months who visited the MCH clinic from 2 September 2018 to 28 September 2018. Outcome measures were socio-demographic, clinical indicators, obstetric indicators, and their relation with overall health-related quality of life score of post-delivery mothers using Short Form Health Survey (SF-36) Version 1.

DETAILED DESCRIPTION:
This cross-sectional study involved women post-delivery to 12 months who visited the Maternal and Child Health (MCH) Clinic of Koshi Hospital, Province 1, Nepal. The study population included the mothers who attended the MCH clinic from post-delivery to 12 months post-delivery. Mothers with psychiatric disorders were excluded from the study population. The investigators used a non-probability purposive sampling technique to select mothers meeting the inclusion criteria. The investigators used Short Form Health Survey (SF-36) Version 1.0 to assess study participants' HRQoL after obtaining permission for Research and Development (RAND). RAND SF-36 was already validated for use in Nepal by Bhandari et al. However, the investigators again pretested the translated Nepali SF-36 among 13 mothers in the MCH Clinic of Tribhuvan University Teaching Hospital. Cronbach's alpha was used to test the reliability, and the reported value was 0.752. Patient participants were involved in the study's pretesting. However, there was no public involvement in the research.

Independent variables: Age of mother, education status, ethnicity, religion, occupation, family income, type of family, family support, parity, number of living children, the desirability of pregnancy, mode of delivery, postpartum duration, place of delivery, and complications in recent delivery.

Dependent variable: Overall health-related quality of life score of post-delivery mothers were used.

Data was collected through face-to-face interviews using the RAND SF-36 Nepali version questionnaire from 2 September 2018 to 28 September 2018. The investigators collected a total of 129 responses. Descriptive statistics, i.e., number, percentage, mean, and standard deviation, were used to describe the demographic and obstetric variables. Mann-Whitney U test was applied to compare postnatal mothers' quality of life in different delivery modes. Similarly, Krushkal-Wallis H and Mann-Whitney U tests were used to examine the difference between the quality of life of postnatal mothers with selected socio-demographic and obstetric variables. Statistical significance was considered with a p-value ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The study population included the mothers who attended the MCH clinic from post-delivery to 12 months post-delivery

Exclusion Criteria:

* Mothers with psychiatric disorders were excluded from the study population.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population included the mothers who attended the MCH clinic from post-delivery to 12 months post-delivery
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2018-08-12 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Quality of Life in Post delivery mothers using RAND 36-Item Short Form Health Survey (SF-36) | 3 months
  Quality of life in Post delivery mothers using RAND 36-Item Short Form Health Survey ranging from 0 to 100, with higher score meaning better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Pratiksha Chapagain, MSc Nursing, Principal Investigator — Maharajgunj Nursing Campus, Tribhuvan University, Institute of Medicine, Kathmandu, Nepal
Locations (1):
- Koshi Hospital, Biratnagar, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Undecided